CLINICAL TRIAL: NCT02514226
Title: Evaluation of Periodontal Treatment in Patients With Bronchiectasis: a Randomized, Single-center,One Year, Parallel Group, Non-inferiority Clinical Study
Brief Title: Evaluation of Periodontal Treatment in Patients With Bronchiectasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Nove de Julho (Other)
Collaborators: InCor Heart Institute (Other); University of Sao Paulo (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Professor of postgraduate program in Biophotonics Applied to Health Sciences, Universidade Nove de Julho, UNINOVE, São Paulo, Brazil, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 44769315.0.0000.5511
Record Dates: First submitted 2015-07-22; First posted 2015-08-03 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Bronchiectasis; Periodontal Disease
Keywords: microbiology; halitosis
MeSH Terms: conditions — Bronchiectasis; Periodontal Diseases; Halitosis | interventions — Periodontal Index; Photochemotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- G1-control group (Placebo Comparator): Arm description: G1 - control group - (n = 30) dental hygiene orientation (DHO) + supragingival treatment + simulation of using photodynamic therapy (PDT).
  In G1, all participants will receive supragingival treatments by an experienced specialist with universal curettes and ultrasound. Supragingival treatment will be performed above the gingival margin. The simulation of using photodynamic therapy (PDT) will be performed with laser turned off. No antibiotics and oral antiseptics will be prescribed.
  Interventions: Procedure: supragingival treatment; Other: dental hygiene orientation
- G2- positive control group (Active Comparator): Arm description: G2 - positive control group (gold standard) - (n = 30) - DHO + periodontal treatment + simulation of using PDT.
  All participants will receive periodontal treatment - scaling and root planning (SRP) by an experienced specialist with universal curetes and ultrasound in a full mouth manner. The simulation of using photodynamic therapy (PDT) will be performed with laser turned off. No antibiotics and oral antiseptics will be prescribed
  Interventions: Procedure: periodontal treatment; Other: dental hygiene orientation
- G3 -experimental active comparator group (Active Comparator): Arm description: G3 - experimental group - (n = 30) DHO +SRP + PDT with methylene blue
  In G3, periodontal treatment and photodynamic therapy (PDT) will be performed. The scaling and root planing will be performed identical as G2. The PDT will be administered in periodontal pockets > 4mm. Methylene blue will be applied in the deep of periodontal pockets. After 5 minutes of application the red laser diode (λ = 660 nm) will be applied with output power of 100 mW with 90 seconds of exposure, i.e. 9J in each point. Applications will be held in six sites around the tooth in all teeth. To finalize, 1 minute of irradiation in scan around each tooth and rinsing with saline solution to remove the photosensitizer
  Interventions: Procedure: periodontal treatment and photodynamic therapy; Other: dental hygiene orientation

INTERVENTIONS:
Procedure: supragingival treatment — In G1, all participants will receive supragingival treatments by an experienced specialist with universal curettes (Hu-Friedy) and ultrasound (Ultra Sound Dabi Atlante - Profi Neo US, Ribeirao Preto, Brazil). Supragingival treatment will be performed above the gingival margin.
  Arms: G1-control group
Procedure: periodontal treatment — All participants receive periodontal treatments by an experienced specialist with universal curettes (Hu-Friedy) and ultrasound (Ultra Sound Dabi Atlante - Profi Neo US, Ribeirao Preto, Brazil) in a full mouth manner.
  Arms: G2- positive control group
Procedure: periodontal treatment and photodynamic therapy — In G3, the periodontal treatment will be performed identical as G2. PDT will be administered in periodontal pockets > 4mm. Methylene blue will be applied in the deep of periodontal pockets. After 5 minutes of application the red laser diode (λ = 660 nm) will be applied with output power of 100 mW (Therapy XT, DMC, São Carlos, Brazil) with 90 seconds of exposure, i.e. 9J in each point. Applications will be held in six sites around the tooth in all teeth. To finalize, 1 minute of irradiation in scan around each tooth and rinsing with saline solution to remove the FS.
  Arms: G3 -experimental active comparator group
Other: dental hygiene orientation — Plaque Control through the use of toothbrush and floss

SUMMARY:
Background: Association between periodontal disease (PD) and chronic obstructive pulmonary disease (COPD) has been widely studied and the aspiration of periodontal pathogens is one of the most accepted causal mechanisms for pulmonary exacerbation. Bronchiectasis is clinically quite similar with COPD, including chronic administration of antibiotics, increased systemic inflammation and relatively similar clinical symptoms, but for the time being; there are no studies that have correlated this condition to PD. This study will evaluate if the scaling and root planning (SRP) associated with photodynamic therapy improves periodontal clinical parameters, halitosis, and the quantity of microorganisms associated with exacerbation of bronchiectasis in saliva, subgingival periodontal microenvironment, sputum and nasal lavage at baseline, after 3 months and one year of SRP. Methods/Design: Ninety patients with chronic periodontal disease and bronchiectasis will be enrolled in the study and they will be treated as follow:G1 control (n = 30) - supragingival scaling (SS) and dental hygiene orientation (DHO); G2 experimental (n = 30) - SRP + DHO; G3- experimental (n = 30) - SRP + PDT + DHO. The quantification of bacterial groups commonly associated with exacerbation of bronchiectasis (P aeruginosa, S. aureus) and periodontal diseases (P. gingivalis), will be evaluated in periodontal pockets, saliva, nasal lavage and sputum by quantitative PCR at baseline 3 months and one year after the SRP. G1 patients will receive SRP upon completion of the investigation. If the mean depth of probing of this group worsen (> 1mm) at 3 months they will be excluded from the study, treated (SRP) and the data will be described. Discussion: The results of this protocol will determine the efficacy of periodontal treatment in decreasing the total amount microorganisms in saliva periodontal pocket, sputum and nasal lavage, the most probable niches of bronchiectasis exacerbation, and reducing local inflammation and halitosis after 3 months and one year. It is expected an higher improvement in all parameters measured over 3 months and 1 year for G3

ELIGIBILITY:
Inclusion Criteria:

* Patients must have > 35 years, both genders, > 10 teeth with chronic moderate generalized periodontal disease , i.e. more than 30% of teeth examined with ≥ 4 mm probing depth.

Exclusion Criteria:

* Exclusion criteria include smokers or former smokers for less than five years, pregnant, people with cystic fibrosis and asthma, phenytoin or cyclosporine users (because they affect periodontal status), decompensated systemic diseases requiring prophylactic antibiotic therapy for periodontal treatment, who used oral antiseptics or anti-inflammatory in the last 3 months, or periodontal treatment performed in the last 6 months.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Microbiological evaluation | 3 months
  Samples will be defrosted and vortexed. DNA extraction will be performed according to manufacturer's instructions. Quantitative PCR of total amount of Bacteria, Archeae, periodontopathogens and Gama-Proteobacteria and Firmicutes groups will be performed with Real-time polymerase chain reaction (PCR)

SECONDARY OUTCOMES:
Halitosis measurements | 3 months
  The air inside the oral cavity will be collected with a syringe and injected into oral ChromaTM, a portable device connected to the computer with captures graph peaks of gas concentration values.

CONTACTS AND LOCATIONS:
Overall Officials: Anna C Horliana, PhD, Principal Investigator — University of Nove de Julho - UniNove
Locations (1):
- InCor Heart Institute, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Romero SS, Pinto EH, Longo PL, Dal Corso S, Lanza FC, Stelmach R, Rached SZ, Lino-Dos-Santos-Franco A, Mayer MP, Bussadori SK, Fernandes KP, Mesquita-Ferrari RA, Horliana AC. Effects of periodontal treatment on exacerbation frequency and lung function in patients with chronic periodontitis: study protocol of a 1-year randomized controlled trial. BMC Pulm Med. 2017 Jan 23;17(1):23. doi: 10.1186/s12890-016-0340-z. PMID 28114928
- [Derived] Pinto EH, Longo PL, de Camargo CC, Dal Corso S, Lanza Fde C, Stelmach R, Athanazio R, Fernandes KP, Mayer MP, Bussadori SK, Mesquita Ferrari RA, Horliana AC. Assessment of the quantity of microorganisms associated with bronchiectasis in saliva, sputum and nasal lavage after periodontal treatment: a study protocol of a randomised controlled trial. BMJ Open. 2016 Apr 15;6(4):e010564. doi: 10.1136/bmjopen-2015-010564. PMID 27084279